CLINICAL TRIAL: NCT04477239
Title: A Randomized, Triple-blind, Placebo-controlled, Clinical Trial on the Diagnostic Performance of Gluten Immunogenic Peptides in the Evaluation of Gluten-free Diet Adherence: the GRRES Study.
Brief Title: Diagnostic Performance of Urinary Gluten Immunogenic Peptides in Monitoring the Adherence to Gluten-free Diet.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Università Politecnica delle Marche (Other)
Responsible Party: Principal Investigator, Carlo Catassi, M.D., Professor, Università Politecnica delle Marche
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Health Services Research
Other Study IDs: GRRES-2020-1551
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Celiac Disease
Keywords: Gluten-free diet; Gluten immunogenic peptides; Gluten contamination; Gluten; Urine
MeSH Terms: conditions — Celiac Disease | interventions — Glutens

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomization will be performed using a random sequence generator to conceal the sequence from the rest of the researchers and to ensure that only the investigator who will manipulate the gluten doses will know the allocation pertaining to each individual. This investigator will not carry out any assessment or any other intervention during the trial period. Until study completion, the enrolled subjects, the clinicians and the person who will perform the statistical analysis will be blinded to the group assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): Oral administration of one capsule of Placebo
  Interventions: Behavioral: Gluten (behaviour); Behavioral: Placebo (behaviour)
- Purified gluten (10 mg) (Active Comparator): Oral administration of capsules containing 10 mg of purified gluten.
  Interventions: Behavioral: Gluten (behaviour); Behavioral: Placebo (behaviour)
- Purified gluten (50 mg) (Active Comparator): Oral administration of capsules containing 50 mg of purified gluten.
  Interventions: Behavioral: Gluten (behaviour); Behavioral: Placebo (behaviour)
- Purified gluten (100 mg) (Active Comparator): Oral administration of capsules containing 100 mg of purified gluten.
  Interventions: Behavioral: Gluten (behaviour); Behavioral: Placebo (behaviour)
- Purified gluten (500 mg) (Active Comparator): Oral administration of capsules containing 500 mg of purified gluten.
  Interventions: Behavioral: Gluten (behaviour); Behavioral: Placebo (behaviour)
- Purified gluten (1000 mg) (Active Comparator): Oral administration of capsules containing 1000 mg of purified gluten.
  Interventions: Behavioral: Gluten (behaviour); Behavioral: Placebo (behaviour)

INTERVENTIONS:
Behavioral: Gluten (behaviour) — Gluten is a protein normally present in the daily diet of healthy volunteers not suffering from gluten related disorders, in far greater quantities (10-20 g/day) than those used in this study (10 mg-1 g/day).
Behavioral: Placebo (behaviour) — Placebo is composed of pregelatinized maize starch Ph.Eur. 97.5%; magnesium stearate Ph.Eur. 1.5%; micronized silica Ph.Eur. 0.5%; Micronized talc Ph.Eur. 0.5% (NOT containing preservatives, colorings, or gluten).

SUMMARY:
The purpose of the GRRES study is to assess the clinical usefulness of urinary gluten immunogenic peptides test as a marker of gluten-free diet adherence using the rapid immunochromatographic assay based on anti-gliadin 33-mer monoclonal antibodies.

DETAILED DESCRIPTION:
A strict and permanent gluten free diet (GFD) is the only effective treatment resulting in full clinical, serological and histological remission, avoiding long-term complications in celiac disease (CD) patients. Gluten immunogenic peptides (GIP) are fragments of gluten proteins resistant to gastrointestinal digestion and detectable in urine after intestinal digestion, providing direct evidence of recent gluten ingestion. A significant variability in the amount of excreted urinary GIP has been reported in individuals administered with similar doses of gluten and, so far, inadequate information is available about the amount of excreted GIP in subjects ingesting traces or low amount of gluten. This is an important issue, as even a strict GFD could be contaminated by traces of gluten, e.g. in wheat starch and processed food. The aim of this study is to assess the clinical usefulness of urinary GIP as a marker of GFD adherence using a rapid immunochromatographic assay based on anti-gliadin 33-mer monoclonal antibodies. This is a prospective, randomized, triple-blind, placebo-controlled, clinical trial. In this study, healthy volunteers following a normal diet will be requested to be on strict GFD for 5 days. On day 4th, participants will be requested to collect a baseline urine sample and in case of a negative GIP test result they will be assigned to ingest a specific dose of purified gluten incorporated in a capsule (0 mg, 10 mg, 50 mg, 100 mg, 500 mg and 1000 mg, according to randomization). Participants will be requested to collect urine samples in a container and take a 5 mL aliquote for the GIP test at the 9th and 24th hour from the time of the administration of the dose. During the collection, volunteers will also be requested to record the volume of the excreted urine and to store the collected urine at 4°C. Urine tubes will be stored at -20°C until the quantitative evaluation of GIP. GIP test will be performed using the rapid immunochromatographic assay based on anti-gliadin 33-mer monoclonal antibodies iVYCHECK GIP Urine™ test (Biomedal, Spain) according to the manufacturer's instructions.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* 20-40 years old
* written informed consent

Exclusion Criteria:

* type 1 diabetes
* chronic or acute inflammatory diseases of the gastrointestinal tract (CD, non-celiac gluten sensitivity, Crohn's disease, ulcerative colitis, food allergy, acute gastroenteritis ≤ 4 weeks prior to the study start)
* pregnancy or lactation
* chronic intake of medications and supplements
* refusal/withdrawal of written informed consent.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Dose-response relationship between the amount of gluten intake and urinary excretion of GIP. | 3 months
  The primary objective of the study is to verify the usefulness of the quantitative GIP assay in urine as biomarker of adherence to the gluten-free diet in terms of dose-response relationship between the amount of ingested gluten and urinary excretion of GIP in a group of healthy volunteers.

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Catassi, MD, MPH, Study Director — Univeristà Politecnica delle Marche, Ancona, Italy; Elena Lionetti, MD, PHD, Principal Investigator — Univeristà Politecnica delle Marche, Ancona, Italy; Simona Gatti, MD, PHD, Study Chair — Univeristà Politecnica delle Marche, Ancona, Italy; Chiara Monachesi, PHD, Study Chair — Univeristà Politecnica delle Marche, Ancona, Italy; Anil K Verma, PHD, Study Chair — Univeristà Politecnica delle Marche, Ancona, Italy
Locations (1):
- University Department of Pediatrics, Ancona, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Moreno ML, Cebolla A, Munoz-Suano A, Carrillo-Carrion C, Comino I, Pizarro A, Leon F, Rodriguez-Herrera A, Sousa C. Detection of gluten immunogenic peptides in the urine of patients with coeliac disease reveals transgressions in the gluten-free diet and incomplete mucosal healing. Gut. 2017 Feb;66(2):250-257. doi: 10.1136/gutjnl-2015-310148. Epub 2015 Nov 25. PMID 26608460
- [Background] Stefanolo JP, Talamo M, Dodds S, de la Paz Temprano M, Costa AF, Moreno ML, Pinto-Sanchez MI, Smecuol E, Vazquez H, Gonzalez A, Niveloni SI, Maurino E, Verdu EF, Bai JC. Real-World Gluten Exposure in Patients With Celiac Disease on Gluten-Free Diets, Determined From Gliadin Immunogenic Peptides in Urine and Fecal Samples. Clin Gastroenterol Hepatol. 2021 Mar;19(3):484-491.e1. doi: 10.1016/j.cgh.2020.03.038. Epub 2020 Mar 23. PMID 32217152
- [Background] Silvester JA, Comino I, Kelly CP, Sousa C, Duerksen DR; DOGGIE BAG Study Group. Most Patients With Celiac Disease on Gluten-Free Diets Consume Measurable Amounts of Gluten. Gastroenterology. 2020 Apr;158(5):1497-1499.e1. doi: 10.1053/j.gastro.2019.12.016. Epub 2019 Dec 19. No abstract available. PMID 31866245
- [Background] Verma AK, Gatti S, Galeazzi T, Monachesi C, Padella L, Baldo GD, Annibali R, Lionetti E, Catassi C. Gluten Contamination in Naturally or Labeled Gluten-Free Products Marketed in Italy. Nutrients. 2017 Feb 7;9(2):115. doi: 10.3390/nu9020115. PMID 28178205
- [Background] Catassi C, Fabiani E, Iacono G, D'Agate C, Francavilla R, Biagi F, Volta U, Accomando S, Picarelli A, De Vitis I, Pianelli G, Gesuita R, Carle F, Mandolesi A, Bearzi I, Fasano A. A prospective, double-blind, placebo-controlled trial to establish a safe gluten threshold for patients with celiac disease. Am J Clin Nutr. 2007 Jan;85(1):160-6. doi: 10.1093/ajcn/85.1.160. PMID 17209192
- [Derived] Monachesi C, Verma AK, Catassi GN, Franceschini E, Gatti S, Gesuita R, Lionetti E, Catassi C. Determination of Urinary Gluten Immunogenic Peptides to Assess Adherence to the Gluten-Free Diet: A Randomized, Double-Blind, Controlled Study. Clin Transl Gastroenterol. 2021 Oct 6;12(10):e00411. doi: 10.14309/ctg.0000000000000411. PMID 34613954